CLINICAL TRIAL: NCT04371458
Title: The Study of Extended Thymectomy and Pleural Reductive Surgery (PRS) With Povidone-iodine Pleural Lavage in Patients With Stage IVA Thymic Malignancies
Brief Title: Thymectomy With and Without Povidone-iodine Pleural Lavage in Stage IVA Thymic Malignancies
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI is not moving forward with study
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000026157
Record Dates: First submitted 2020-04-28; First posted 2020-05-01 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Stage IVA Thymoma
Keywords: Intra-Pleural Providone-Iodine
MeSH Terms: conditions — Thymoma

STUDY DESIGN:
Intervention Model Description: Intraoperative providone-iodine lavage during resection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoperative providone-iodine lavage (Experimental): Intraoperative providone-iodine lavage during resection
  Interventions: Drug: Intraoperative providone-iodine lavage

INTERVENTIONS:
Drug: Intraoperative providone-iodine lavage — Intraoperative providone-iodine lavage during resection

SUMMARY:
To evaluate whether intraoperative pleural lavage with providone-iodine following complete resection and pleural reductive surgery for stage IVA thymoma reduces recurrent rates compared to surgery without providone-iodine lavage

DETAILED DESCRIPTION:
Following the surgical portion of the procedure, assuming frozen section confirms the suspected diagnosis, pleural lavage using 10% povidone-iodine (warmed to normothermic 37°C) will begin. The 10% povidone-iodine is mixed with sterile water with a dilution of 1/10. A total of 6-14 liters of solution will be prepared in advance of the procedure, pending the size of the patient's chest cavity. The warmed PVP-I will be instilled into the chest cavity to a volume that fills involved thoracic cavity or cavities. Once filled, the solution will be allowed to dwell for 15 minutes. At the conclusion of the 15 minutes, the PVP-I solution will be suctioned out of the chest. This process will be repeated for a total of three dwell sessions.

At the conclusion of the PVP-I lavage, chest tubes should be placed in the chest cavity to re-expand the lung adequately. Chest tube management will be at the discretion of the individual thoracic surgeons, including suction vs water seal and plan for removal.

An honest attempt to maintain the management according to the study protocol will be made. However, if it deemed inappropriate for that patient due to clinical signs, symptoms, or anticipated problems, the surgical team can make whatever changes are deemed necessary. The reason for the deviation must be documented. This patient's data will continue to be collected and analyzed on an intent-to-treat basis for the primary, secondary and tertiary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group - PS 0 or 1
* Patients with a histologic diagnosis of thymic epithelial tumor (thymoma WHO type A, AB, B1, B2, B3; or thymic carcinoma) who in the opinion of the attending thoracic surgeon can technically receive a macroscopic complete resection of pleural nodules. This histologic diagnosis can be obtained either preoperatively, or based on frozen section intra-operatively.
* Signed informed consent form
* Completely resectable burden of disease
* No evidence of distant organ metastasis except resectable pulmonary parenchymal nodules and intrathoracic lymph node metastasis as evidenced by CT chest, physical examination, and any other indicated studies
* Medically suitability for resection as determined by the operating surgeon
* Women of childbearing potential (WOCBP) must have a negative urinary pregnancy test pre-operatively

Exclusion Criteria:

* Patients with active invasive cancers, other than thymoma, that requires treatment, except non-melanomatous skin cancer, superficial bladder cancer or cervical cancer and early stage prostate cancer.
* If frozen section reveals a diagnosis other than thymoma or thymic carcinoma, the patient will be removed from protocol and the providone-iodine lavage will not be performed.
* Hyperthyroidism or Radioisotope treatment for thyroid disease.
* Radiographic evidence of disease beyond the primary site and pleural space
* History of pulmonary resection more than lobectomy. (regardless of laterality)
* Pregnant or lactating patients
* Patients with iodine allergy
* Patients who have severe liver disease including cirrhosis, grade III-IV elevations in liver function studies, or bilirubin in excess of 1.5 mg/decilitre
* Pulmonary nodules or visceral nodules requiring pulmonary resection sacrificing more than half of ipsilateral lung parenchyma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 5 years
  Progression free survival as compared to that of matched patients in a prospectively enrolled international database of thymic malignancies (ITMIG)

SECONDARY OUTCOMES:
Pleural recurrence | 5 years
  Pleural recurrence will be assessed with CT scans of the chest every 6 months starting 6 months after the index operation and continuing for 3 years. After 3 years, if no recurrence has been identified yet, patients will get CT scans of the chest on an annual basis.
Overall survival | 5 years
  Overall survival will be assessed by regular patient evaluations, which will correspond with the CT scans of the chest. If a patient expires, date and cause of death will be recorded. Causes related to thymic malignancy will be differentiated from other causes of mortality to arrive at disease-specific survival and all-cause overall survival.
Patient and disease characteristics | 5 years
  Identification of patient and disease characteristics associated with improved responses to providone-iodine lavage.
  Variables examined will include demographic data such as age, sex and comorbidities. Additional data evaluated will include specific aspects of the primary thymic tumor such as burden of thoracic disease (confined to mediastinum, extension into ipsilateral pleura, burden of disease in pleura), and pathology characteristics (WHO Type, level of differentiation).

IPD SHARING:
Plan to Share IPD: No